CLINICAL TRIAL: NCT00643825
Title: Randomized Multicentric Phase II Study of Prolonged Adjuvant Temozolomide or "Stop and Go" in Glioblastoma Patients: The PATSGO Study
Brief Title: Prolonged Adjuvant Temozolomide vs "Stop & Go" in Glioblastoma Patients
Acronym: PATSGO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Prof Baurain J-Fr, Cliniques universitaires Saint-Luc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL-ONCO 06-004
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Glioblastoma
Keywords: Temozolomide; Phase II; Chemotherapy; Glioblastoma; Progression-free Survival
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: prolonged adj TMZ (Active Comparator)
  Interventions: Drug: Temozolomide
- B : Stop and Go (Other): Rechallenging patients with TMZ at relapse
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Capsules 5,10,20,100,250 mg 200mg/m2/day , 5days per 28 till PD
  Other Names: TEMODAR, TEMODAL
  Arms: A: prolonged adj TMZ
Drug: Temozolomide — Observation till Progression then rechallenging with TMZ
  Other Names: TEMODAR, TEMODAL
  Arms: B : Stop and Go

SUMMARY:
This study will test the hypothesis that prolonged adjuvant Temozolomide (TMZ) may delay relapses in patients with glioblastoma compared to the standard care consisting in observation with brain MRI every 3 months and rechallenging with TMZ at relapse (Stop and Go arm).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed diagnosis of GBM
2. Availability of pre-treatment GBM tissue to determine the activation status of MGMT gene is not mandatory but strongly recommended
3. Patients must have received radiation and TMZ for 6 weeks followed by 6 months of TMZ. Randomization should be performed within the 6 weeks after the last chemotherapy.
4. A brain MRI with or without a PET-Scan-methionine must be performed before enrolment.
5. Age ≥ 18 years
6. Karnofsky Performance status ≥ 60
7. Normal haematological functions: ANC ≥ 1.5 x 109cells/l, platelets ≥ 100 x 109 cells/l
8. Normal liver function: total bilirubin < 1.5 x ULN, alkaline phosphatase and transaminases (ASAT/ALAT) < 2.5 times the upper limit of the normal range
9. Serum creatinine < 1.5 x ULN
10. Clinically normal cardiac function without history of ischemic heart disease in the past 12 months. Absence of cardiac insufficiency NYHA grade III and IV, instable angina, arrhythmia
11. No previous or current malignancy (except treated basal or squamous cell skin carcinoma, cervix cancer or in situ carcinoma of the breast).
12. All patients (male and female) with reproductive potential must use effective contraception. Females must have a negative serum pregnancy test at entry to study.
13. Signed informed consent from the patient or legal representative must be obtained.

Exclusion Criteria:

All non inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
to determine whether prolonged administration of Temozolomide in glioblastoma patients increase their progression-free and overall survival at 6 months | 36 months

SECONDARY OUTCOMES:
safety and adverse event profile of prolonged adjuvant Temozolomide | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Baurain, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Europe, Belgium